# **COVER PAGE**

### **Informed Consent Form**

OFFICIAL TITLE: Evaluation of computed tomography and magnetic diffusion resonance imaging in the preoperative staging of colon cancer

BRIEF TITLE: CT and MRI in Preoperative Colon Cancer Staging

**UNIQUE PROTOCOL ID:** CTMR **DOCUMENT DATE:** January 2023

### **Principal Investigator:**

Effrosyni Bompou, MSc Telephone: 00302413501000 Email: feybobou@hotmail.com

### **Sub-Investigators:**

Ioannis Baloyiannis Aikaterini Vassiou

### **Study Director**

George Tzovaras, Professor of General Surgery

Telephone: 00302413502804 Email: gtzovaras@hotmail.com

> Department of Surgery University Hospital of Larissa Mezourlo 41110 Larissa Greece

## UNIVERSITY OF THESSALY, DEPARTMENT OF

UNIVERSITY GENERAL HOSPITAL OF LARISSA Mezourlo, 41110, Larissa



**Director: Professor Zacharoulis Dimitrios** A 'Building, 2nd Floor, P.G.N. Of Larissa



### UNIVERSITY OF THESSALY, FACULTY OF MEDICINE

UNIVERSITY HOSPITAL OF LARISSA Mezourlo, 41110, Larissa GREECE

#### GENERAL SURGERY DPT

Chairman: Prof. Zacharoulis Dimitrios A 'Wing, 2nd Floor, University Hospital of Larissa

### **Research Protocol**:

# Evaluation of computed tomography and magnetic diffusion resonance imaging in the preoperative staging of colon cancer

The objective of this study is the evaluation of different imaging methods for the optimal preoperative staging of colon cancer patients. Imaging findings will be compared with the histopathologic results of the specimen following surgical resection. The study protocol is designed as a prospective study.

### 1. Procedure

The patient will be admitted to the surgical department according to the predetermined procedure. All the necessary preoperative imaging and laboratory examinations will be performed. A multidisciplinary oncology board will follow to determine the optimal treatment. Following this, the patient will be submitted to the optimal operation for him / her to treat his / her condition. Postoperatively the patient will be monitored in the surgical department according to the existing protocols and guidelines.

### 2. Dangers

The risks are related to the possible postoperative complications from the operation.

### 3. Expected benefits

The research will result to the publication of data - results. Your participation in the protocol implies that you agree with future publication of results, provided that the information will be anonymous, and the names of the participants will not be disclosed. The data that will be collected will be encoded with a number, so that your name will not appear anywhere.

### 4. Information

Do not hesitate to ask questions regarding the purpose or the process of the protocol. If you have any doubts or questions, please ask us to give you clarifications.

### 5. Participation

Your participation in the protocol is voluntary. You are free to disagree or cancel your participation whenever you wish.

### 6. Informed consent

| | I have | read | this | form | and | I | understand | the | processes | that | I | will | follow. | I | agree | to |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| par | ticipate | in the | rese | arch p | oroto | co | 1. | | | | | | | | | |

| Date:/ | <u></u> |
|--------|----------------|
| Partic | ipant Name and |
| Signa | ture |

Investigator Signature

Principal Investigator: Effrosyni Bompou, MSc Telephone: 00302413501000 Email: feybobou@hotmail.com

### **Study Director:**

George Tzovaras, Professor of General Surgery Telephone: 00302413502804 Email: gtzovaras@hotmail.com